CLINICAL TRIAL: NCT04566510
Title: Impact of Long-lasting Insecticidal Nets (LLINs) Treated With Pyrethroid Plus Pyriproxyfen vs LLINs Treated With Pyrethroid Plus Piperonyl Butoxide on Malaria Incidence in Uganda: a Cluster-randomised Trial
Brief Title: LLIN Evaluation in Uganda Project
Acronym: LLINEUP2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LLINEUP2; U19AI089674 (NIH)
Record Dates: First submitted 2020-09-22; First posted 2020-09-28 (Actual); Results first posted 2024-11-14 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Malaria
Keywords: long-lasting insecticidal net; pyriproxyfen; piperonyl butoxide; alpha-cypermethrin; deltamethrin
MeSH Terms: conditions — Malaria | interventions — cypermethrin; pyriproxyfen; decamethrin; Piperonyl Butoxide

STUDY DESIGN:
Intervention Model Description: cluster-randomised trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Royal Guard (Experimental): alpha-cypermethrin + pyriproxyfen (PPF)
  Interventions: Other: long lasting insecticidal nets with alpha-cypermethrin + pyriproxyfen (PPF LLIN, Royal Guard)); Behavioral: Social behaviour change communication
- PermaNet 3.0 (Active Comparator): deltamethrin + piperonyl butoxide (PBO)
  Interventions: Other: long lasting insecticidal nets with deltamethrin + piperonyl butoxide (PBO LLIN, PermaNet 3.0)); Behavioral: Social behaviour change communication

INTERVENTIONS:
Other: long lasting insecticidal nets with alpha-cypermethrin + pyriproxyfen (PPF LLIN, Royal Guard)) — Next-generation bed net combining insecticides with different modes of action
  Arms: Royal Guard
Other: long lasting insecticidal nets with deltamethrin + piperonyl butoxide (PBO LLIN, PermaNet 3.0)) — Next-generation bed net combining an insecticide with a synergist
  Arms: PermaNet 3.0
Behavioral: Social behaviour change communication — SBCC activities will use digital and other platforms, similar to those used for the COVID-19 response, including the following: (1) LLIN launch on television and radio; (2) regional advocacy meetings on Zoom; (3) mass media platforms (for advertisements, mini skits, DJ mentions, radio spots, interactive talks); (4) social media platforms; (5) VHTs; (6) operation hotlines and toll-free call centres; (7) community mobilisation (megaphones); and (8) use of appropriate information, education, and communication materials. Communication will include messages about COVID-19, malaria, and use, care, repair and repurposing of LLINs.

SUMMARY:
In Uganda, the National Malaria Control Division (NMCD) and implementing partners plan to deliver long-lasting insecticidal nets (LLINs) nationwide in 2020-21, through a mass distribution campaign supported by generous contributions from international donors. LLINs will be distributed free-of-charge to all Ugandan households, aiming to achieve universal coverage. The Against Malaria Foundation has agreed to provide LLINs treated with a pyrethroid insecticide plus pyriproxyfen (PPF) (Royal Guard, Disease Control Technology) and LLINs treated with a pyrethroid insecticide plus piperonyl butoxide (PBO) (PermaNet 3.0, Vestergaard), presenting an opportunity to rigorously evaluate and compare these two LLINs at scale across Uganda. In collaboration with the MOH, the investigators propose to embed a cluster-randomised trial to compare the impact of LLINs with PPF to LLINs with PBO into Uganda's 2020 LLIN distribution campaign. The primary objective of the study is: To evaluate the impact of LLINs treated with a pyrethroid insecticide plus pyriproxyfen (PPF LLINs), as compared to LLINs treated with a pyrethroid plus piperonyl butoxide (PBO LLINs), on malaria incidence in Uganda. The study will test the hypothesis that malaria incidence will be lower in intervention clusters (randomised to receive PPF LLINs) than in control clusters (randomised to receive PBO LLINs).

DETAILED DESCRIPTION:
This rigorous, cluster-randomised trial will evaluate the impact of long-lasting insecticidal nets (LLINs) distributed in Uganda through the 2020-21 national universal coverage campaign. A cluster has been defined as the catchment area of a Malaria Reference Centre (MRC). A total of 64 clusters have been included in the study, covering 32 high malaria burden districts in Uganda where IRS is not being implemented. Clusters have been randomised in a 1:1 ratio in blocks of two by district to receive one of two types of LLINs: (1) pyriproxyfen (PPF) LLINs (Royal Guard) [n=32] and (2) piperonyl butoxide (PBO) LLINs (PermaNet 3.0) [n=32].

The intervention, including delivery of the LLINs and social and behaviour change communication (SBCC), will be led by the Ugandan National Malaria Control Division (NMCD) and other stakeholders. Currently, LLINs are scheduled to be delivered in the study areas from October 2020 to January 2021. The evaluation will include health facility surveillance at the MRCs to generate continuous estimates of malaria incidence for each MRC catchment area, cross-sectional community surveys at baseline (if additional resources are available), and at 12- and 24-months after LLIN distribution to gather information on net survivorship and use, and parasite prevalence in children 2-10 years of age, entomology surveys, and assessment of net durability and efficacy. The primary outcome of the trial will be malaria incidence as estimated using the health facility surveillance.

For each cluster the study will use a 'fried egg' approach for delivering the intervention ('egg white') and measuring our outcomes ('egg yolk'). The 'white' of the egg will include one sub-county per cluster, where the MRC is located. PPF LLINs and PBO LLINs will be distributed to the designated sub-county, as allocated in the randomisation. The 'yolk' of the egg will be the catchment area directly surrounding each MRC, where care-seeking at the MRC is expected to be high (i.e. if someone within the catchment area develops malaria, they are likely to seek care at the MRC). To determine the population of the MRC catchment areas, and to generate a sampling frame for the community surveys, the investigators will do the following: (1) define the catchment area of each MRC before the onset of the trial using data on village of residence from patients attending the MRCs, (2) map and enumerate all households within the MRC catchment areas before the 12-month community survey, and (3) conduct a census survey within each MRC catchment area to generate an accurate estimate of the study population in which study outcomes will be measured concurrently with the 12-month community survey.

ELIGIBILITY:
A) Primary outcome: All patients who present to the outpatient departments of the MRCs

B) Community surveys for secondary outcomes:

Inclusion Criteria:

* At least one adult aged 18 years or older present
* Adult is a usual resident who slept in the sampled household on the night before the survey
* Agreement of the adult resident to provide informed consent for the household survey

Exclusion Criteria:

* Dwelling destroyed or not found
* Household vacant
* No adult resident home on more than 3 occasions

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 32895 (Actual)
Dates: Start 2020-10-17 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Staedke, MD, PhD, Principal Investigator — London School of Hygiene and Tropical Medicine; Moses Kamya, MBChB, MMed, PhD, Principal Investigator — Infectious Diseases Research Collaboration
Locations (1):
- Infectious Diseases Research Collaboration, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gonahasa S, Namuganga JF, Nassali MJ, Maiteki-Sebuguzi C, Nabende I, Epstein A, Snyman K, Nankabirwa JI, Opigo J, Donnelly MJ, Dorsey G, Kamya MR, Staedke SG. LLIN Evaluation in Uganda Project (LLINEUP2) - Effect of long-lasting insecticidal nets (LLINs) treated with pyrethroid plus pyriproxyfen vs LLINs treated with pyrethroid plus piperonyl butoxide in Uganda: A cluster-randomised trial. PLOS Glob Public Health. 2025 Feb 26;5(2):e0003558. doi: 10.1371/journal.pgph.0003558. eCollection 2025. PMID 40009611

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Households from each of the 64 clusters was randomly selected for participation in each of the community surveys. Within each cluster (MRC target area), households were randomly sampled from a list of households enumerated by the study team, until 50 households with children aged 2-10 years were sampled per cluster.
Pre-assignment Details: Only participants in the MRC target areas who participated in cross sectional surveys were considered enrolled while all other persons living in the target areas were not enrolled.
Units Other Than Participants: MRC target area
Period: 12 Month Cross Sectional Survey
Arm/Group | Royal Guard | PermaNet 3.0
Started (All residents from selected households that provided informed consent were enrolled.) | 7940; 32 MRC target area | 8249; 32 MRC target area
Completed | 7940; 32 MRC target area | 8249; 32 MRC target area
Not Completed | 0; 0 MRC target area | 0; 0 MRC target area
Period: 24 Month Cross Sectional Period
Arm/Group | Royal Guard | PermaNet 3.0
Started (All residents from selected households that provided informed consent were enrolled.) | 8306; 32 MRC target area | 8400; 32 MRC target area
Completed | 8306; 32 MRC target area | 8400; 32 MRC target area
Not Completed | 0; 0 MRC target area | 0; 0 MRC target area

BASELINE CHARACTERISTICS:
Population: Estimated number of persons living in 64 MRC target areas used in primary outcome; only persons enrolled in cross-sectional surveys were consented and enrolled and included within this estimated number
Groups:
- Total: Total of all reporting groups
Arm/Group | Royal Guard | PermaNet 3.0 | Total
Number analyzed (Participants) | 92648 | 99132 | 191780
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.7 (17.6) | 19.9 (17.3) | 19.8 (17.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46324 | 49566 | 95890
  Male | 46324 | 49566 | 95890
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 92648 | 99132 | 191780
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Incidence of malaria in residence of all ages from MRC target areas [Number; unit: episodes of malaria over 3 months] | 15621 | 16763 | 32384

OUTCOME MEASURES:

1. Primary Outcome: Malaria Incidence
Description: Number of cases of laboratory-confirmed malaria diagnosed at the MRC among patients residing in the catchment areas per unit time/the population of the catchment areas
Time Frame: 24 months following LLIN distribution
Population: estimated number of residents of all ages from MRC target areas; these estimates came from routine surveillance data that did not involve consent or enrollment
Measure: Number; unit: episodes of malaria over 24 months
Arm/Group | Royal Guard | PermaNet 3.0
Number analyzed (Participants) | 96360 | 103106
episodes of malaria over 24 months | 90466 | 95898

2. Secondary Outcome: Prevalence of Parasitaemia
Description: Proportion of children aged 2-10 years at the time of cross-sectional surveys with blood smears positive for parasites by microscopy
Time Frame: 12 months following LLIN distribution
Population: children 2-10 years of age enrolled in cross-sectional surveys
Measure: Number; unit: participants with parasitemia
Arm/Group | Royal Guard | PermaNet 3.0
Number analyzed (Participants) | 2482 | 2411
participants with parasitemia | 654 | 521

3. Secondary Outcome: Prevalence of Parasitaemia
Description: Proportion children aged 2-10 years at the time of cross-sectional surveys with blood smears positive for parasites by microscopy
Time Frame: 24 months following LLIN distribution
Population: children 2-10 years of age enrolled in cross-sectional surveys
Measure: Number; unit: participants with parasitemia
Arm/Group | Royal Guard | PermaNet 3.0
Number analyzed (Participants) | 2208 | 2311
participants with parasitemia | 651 | 602

4. Secondary Outcome: Prevalence of Anaemia
Description: Proportion of children aged 2-4 years with haemoglobin < 11 g/dL at the time of cross-sectional surveys
Time Frame: 12 months following LLIN distribution
Population: children 2-4 years of age enrolled in cross-sectional surveys
Measure: Number; unit: participants with hemoglobin <11g/dL
Arm/Group | Royal Guard | PermaNet 3.0
Number analyzed (Participants) | 1022 | 1065
participants with hemoglobin <11g/dL | 347 | 385

5. Secondary Outcome: Prevalence of Anaemia
Description: Proportion of children aged 2-4 years with haemoglobin < 11 g/dL at the time of cross-sectional surveys
Time Frame: 24 months following LLIN distribution
Population: children 2-4 years of age enrolled in cross-sectional surveys
Measure: Number; unit: participants with hemoglobin <11g/dL
Arm/Group | Royal Guard | PermaNet 3.0
Number analyzed (Participants) | 937 | 971
participants with hemoglobin <11g/dL | 178 | 191

6. Secondary Outcome: Proportion of Households That Owned at Least One LLIN
Description: Proportion of households with at least one LLIN at the time of cross-sectional surveys
Time Frame: 12 months following LLIN distribution
Population: households enrolled in 12 month cross-sectional surveys
Measure: Number; unit: households with at least 1 LLIN
Units Other Than Participants: households
Arm/Group | Royal Guard | PermaNet 3.0
Number analyzed (Participants) | 7940 | 8249
Number analyzed (households) | 1747 | 1771
households with at least 1 LLIN | 1571 | 1628

7. Secondary Outcome: Proportion of Households That Owned at Least One LLIN
Description: Proportion of households with at least one LLIN at the time of cross-sectional surveys
Time Frame: 24 months following LLIN distribution
Population: households enrolled in 24 month cross-sectional surveys
Measure: Number; unit: households with at least 1 LLIN
Units Other Than Participants: households
Arm/Group | Royal Guard | PermaNet 3.0
Number analyzed (Participants) | 8306 | 8400
Number analyzed (households) | 1682 | 1690
households with at least 1 LLIN | 1345 | 1384

8. Secondary Outcome: Proportion of Households That Owned at Least One LLIN for Every Two Occupants
Description: Proportion of households with at least one LLIN per every two occupants at the time of cross-sectional surveys
Time Frame: 12 months following LLIN distribution
Population: households enrolled in 12 month cross-sectional surveys
Measure: Number; unit: households with at least 1 LLIN/2persons
Units Other Than Participants: households
Arm/Group | Royal Guard | PermaNet 3.0
Number analyzed (Participants) | 7940 | 8249
Number analyzed (households) | 1747 | 1771
households with at least 1 LLIN/2persons | 987 | 1060

9. Secondary Outcome: Proportion of Households That Owned at Least One LLIN for Every Two Occupants
Description: Proportion of households with at least one LLIN per every two occupants at the time of cross-sectional surveys
Time Frame: 24 months following LLIN distribution
Population: households enrolled in 24 month cross-sectional surveys
Measure: Number; unit: households with at least 1LLIN/2persons
Units Other Than Participants: households
Arm/Group | Royal Guard | PermaNet 3.0
Number analyzed (Participants) | 8306 | 8400
Number analyzed (households) | 1682 | 1690
households with at least 1LLIN/2persons | 650 | 695

10. Secondary Outcome: Proportion of Household Residents Who Slept Under an LLIN the Previous Night
Description: Proportion of households residents who report sleeping under LLIN the previous night at the time of cross-sectional surveys
Time Frame: 12 months following LLIN distribution
Population: household residents enrolled in 12 month cross-sectional surveys
Measure: Number; unit: residents reported sleeping under LLIN
Arm/Group | Royal Guard | PermaNet 3.0
Number analyzed (Participants) | 7940 | 8249
residents reported sleeping under LLIN | 6045 | 6121

11. Secondary Outcome: Proportion of Household Residents Who Slept Under an LLIN the Previous Night
Description: as for outcome 10
Time Frame: 24 months following LLIN distribution
Population: household residents enrolled in 24 month cross-sectional surveys
Measure: Number; unit: residents reporting sleeping under LLIN
Arm/Group | Royal Guard | PermaNet 3.0
Number analyzed (Participants) | 8306 | 8400
residents reporting sleeping under LLIN | 5117 | 5341

ADVERSE EVENTS:
Description: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Arm/Group | Royal Guard | PermaNet 3.0
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2023-10-17): https://cdn.clinicaltrials.gov/large-docs/10/NCT04566510/Prot_000.pdf
  • Statistical Analysis Plan (2023-01-25): https://cdn.clinicaltrials.gov/large-docs/10/NCT04566510/SAP_001.pdf